CLINICAL TRIAL: NCT02272751
Title: A Comparison of Exercise Training With Relaxation Intervention in Lymphoma Patients Post-chemotherapy.
Brief Title: Relaxation and Exercise In Lymphoma Patients
Acronym: REIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13.0108
Record Dates: First submitted 2014-10-16; First posted 2014-10-23 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Lymphoma; Quality of Life
Keywords: cancer survivorship; exercise; relaxation; mindfulness
MeSH Terms: conditions — Lymphoma; Motor Activity | interventions — Exercise; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Intervention (Experimental): Subjects allocated to the Exercise arm will aim to undertake a personal prescribed home exercise programme for half an hour three times a week.
  Exercises will be progressed at 6 weeks as subjects progress. All exercise sessions will be documented in the logbooks provided.
  Outcome measures will be assessed at baseline, mid-way (6 weeks) and at the end of intervention (12 weeks).
  Interventions: Behavioral: Exercise
- Relaxation Intervention (Experimental): Subjects allocated to the Relaxation arm will aim to undertake a guided relaxation programme on a CD for half an hour three times a week.
  All relaxation sessions will be documented in the logbooks provided. Outcome measures will be assessed at baseline, mid-way (6 weeks) and at the end of intervention (12 weeks).
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Exercise — The Exercise intervention will consist of aerobic activity followed by upper and lower limb resistance training using Therabands and some core exercises.
  Other Names: Exercise Training
  Arms: Exercise Intervention
Behavioral: Relaxation — The Relaxation intervention will consist of a chair-based program incorporating breathing exercises, meditation, visualisation and progressive muscle relaxation.
  Other Names: Mindfulness
  Arms: Relaxation Intervention

SUMMARY:
This study will aim to compare the effects of an Exercise programme and a Relaxation Intervention in lymphoma patients in remission post-chemotherapy on quality of life, cardiovascular fitness, exercise tolerance, muscle strength, psychological status, social well-being and biological markers.

Subjects will be recruited from a specialist lymphoma clinic in South West London and randomly allocated to an exercise or a relaxation home programme. The study aims to determine the more effective intervention of the two in relation to the outcome measures.

The investigators anticipate that the interventions will result in less adverse events and improved quality of life and physical fitness, and subjects will require less medication, less counseling and cancer nurse specialist care, leading to leading to a reduction in hospital and surgery attendances.

DETAILED DESCRIPTION:
Significant improvements have been made in the survival rates in cancer patients. Due to factors such as screening and earlier detection of cancer and advances in treatment, cancer today is a curable disease for many. However, cancer survivors are at a significantly increased risk of morbidity and adverse effects due to treatment exposures. Commonly reported consequences of cancer treatment include fatigue, pain, depression, anxiety, reduced performance status and decreased quality of life Hence cancer today is considered more as a chronic illness, and there is increasing research being carried out on cancer survivorship and recommendations for survivorship care pathways to include interventions to enhance both physical and psychosocial functioning in cancer survivors.

Previous studies have demonstrated that both exercise and interventions such as relaxation have a positive effect on both physical and psychosocial complaints of cancer survivors. These interventions are carried out in different ways, have different requirements and perceptions of the two can also be very different. No trial to date has been carried out comparing the effects of these interventions on the quality of life in cancer survivors. Furthermore, majority of the above research has been carried out on the most prevalent cancers including breast cancer, prostate cancer and colorectal cancer, and several authors have called for future research to focus on other understudied survivor groups, including haematologic cancer sites. This study aims to compare the effect of exercise and relaxation interventions on quality of life in lymphoma survivors.

The aim of the present study is to compare the effects of an Exercise Intervention Program with a Relaxation Intervention in a sample of lymphoma patients in remission post-chemotherapy.

Eligible subjects will be randomised to one of two arms - either an exercise or a relaxation arm. Both arms comprise of a home programme of their intervention (either exercise or relaxation) for half an hour, carried out three times a week. Subjects are assessed using the primary and secondary outcome measures at baseline, midway (6 weeks) and at the end of the intervention (12 weeks). It is hypothesised that a 12 week training programme of both exercise and relaxation would improve the quality of life of lymphoma survivors, however the exercise programme would result in a significantly greater improvement than relaxation. The null hypothesis would state that there would be no significant difference between exercise or relaxation groups following a 12 week training programme in lymphoma survivors.

The aims of the study are as follows:

Primary aim

To compare the effectiveness of Exercise with Relaxation in the improvement of overall wellbeing and quality of life using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30).

Secondary aims

To determine whether these interventions result in:

* Improved cardio-respiratory fitness (resting HR and BP) and pulmonary function (spirometry)
* Improved fitness and exercise tolerance using the 6 Minute Walk Test
* Improved emotional and functional confidence as measured by the Health related quality of life questionnaire Functional Assessment of Cancer Therapy Lymphoma version (FACT-Lym)
* Decreased anxiety and depression levels using the Hospital Anxiety and Depression Scale (HADS)
* Changes in haematology (haemoglobin, immunoglobulins, white count) and biochemical (serum albumin, corrected calcium, creatinine) parameters
* Compare the results of the above outcome measures between the two interventions
* Analyse subject perceptions of interventions in focus groups

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed lymphoma in remission post-chemotherapy
2. Age 18 years or older
3. Ability to give informed consent
4. Good Performance status (ECOG 0-2)
5. Clinically able to carry out exercise training programme on a regular basis

Exclusion Criteria:

1. Patients with progressive disease
2. Poor performance status (ECOG status 3 or more)
3. Abnormal resting ECG unexplained by further cardiological investigations
4. Pregnancy
5. Difficulty breathing at rest
6. Persistent cough, fever or illness
7. Cognitive impairment sufficient to limit ability to perform quality of life questionnaires or understand instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline, 6 weeks and 12 weeks
  The EORTC-QLQ-C30 is a self-administered questionnaire which assesses aspects of function, symptoms, and global health and QOL in samples of cancer patients. It has been demonstrated to be a valid and reliable tool in the literature, takes approximately eleven minutes to complete and most subjects require no assistance.

SECONDARY OUTCOMES:
Change in Six Minute Walk Test distance and Heart Rate | Baseline, 6 weeks and 12 weeks
  The Six Minute Walk Test (6MWT) is a valid and reliable tool used in a variety of clinical settings, and validated for use with cancer patients. The patient is read out a set of standardised instructions to walk around a measured distance continuously as fast as they can for six minutes. Following this, the distance covered is measured and recorded, as well as their Heart Rate, Saturations, Rate of Perceived Exertion and Dyspnoea (using Borg scales) are recorded.
  This test gives an indication of general fitness and overall function.
Change in Grip Strength | Baseline, 6 weeks and 12 weeks
  Grip strength will be determined using hand-held dynamometry following a set of standardised guidelines. This is a common method that is used extensively to assess general strength characteristics.
Change in Spirometry values | Baseline, 6 weeks and 12 weeks
  Measures of pulmonary capacity and function including Forced Vital Capacity (FVC), Forced Expiratory Volume in one second (FEV1), Forced Expiratory Ratio (FER) and Peak Expiratory Flow (PEF) will be taken via microspirometry.
Change in FACT-Lym Questionnaire | Baseline, 6 weeks and 12 weeks
  The Functional Assessment of Chronic Illness questionnaires, have been validated in studies of cancer management and are designed to encompass the whole range of psychosocial factors. Here, the lymphoma-specific (FACT-Lym) self-administered questionaire will be used.
Change in Hospital Anxiety and Depression Scale | Baseline, 6 weeks and 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a valid tool for the identification of psychiatric complications of cancer such as depression, anxiety or distress in cancer settings. It is a self-administered questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pettengell, MBChB PhD, Principal Investigator — St George's, University of London; Ahmed Younis, PhD, Study Director — St George's, University of London
Locations (1):
- Haematology and Oncology Outpatient Clinic, St. George's Hospital, Blackshaw Road, Tooting, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be submitted for publication, undecided re: individual participant data

REFERENCES:
- [Derived] Hathiramani S, Pettengell R, Moir H, Younis A. Relaxation versus exercise for improved quality of life in lymphoma survivors-a randomised controlled trial. J Cancer Surviv. 2021 Jun;15(3):470-480. doi: 10.1007/s11764-020-00941-4. Epub 2020 Sep 28. PMID 32986231
- [Derived] Hathiramani S, Pettengell R, Moir H, Younis A. Relaxation and exercise in lymphoma survivors (REIL study): a randomised clinical trial protocol. BMC Sports Sci Med Rehabil. 2019 Aug 16;11:17. doi: 10.1186/s13102-019-0127-7. eCollection 2019. PMID 31428434